CLINICAL TRIAL: NCT06957613
Title: A Prospective Follow-up Assessment in Bad Segeberg With Patients Undergoing Recanalization of Coronary Lesions With Chronic Total Occlusion
Brief Title: The Prospective Segeberg Registry for Coronary Chronic Total Occlusions (CTO)
Acronym: CTO Registry
Status: Recruiting | Type: Observational
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SK 112 - 168/11
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Chronic Total Occlusions
Keywords: Chronic Total Occlusion
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Coronary Chronic Total Occlusions: Patients undergoing Recanalization for Coronary Chronic Total Occlusions
  Interventions: Procedure: Revascularization/Conservative management

INTERVENTIONS:
Procedure: Revascularization/Conservative management — Percutaneous Transluminal Angioplasty of Coronary Chronic Total Occlusions via Dedicated Drug Eluting Stents and/or Balloons.

SUMMARY:
A Prospective Follow-up Assessment in Bad Segeberg with Patients undergoing Recanalization for Coronary Chronic Total Occlusion Lesion/s

DETAILED DESCRIPTION:
A prospective single center registry including all patients treated for Chronic Total Occlusion Coronary Lesion/s at the Heart Center, Bad Segeberg, Germany. Patients undergo a routine clinical follow-up schedule, including a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary chronic total occlusions undergoing recanalization via percutaneous coronary interventions

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary chronic total occlusions undergoing recanalization vie percutaneous coronary interventions
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of in-hospital and long-term cardiovascular adverse events in percent | 2 years
  Peri-procedural events and in-hospital cardiovascular events and long-term cardiovascular events (bleeding, peripheral and coronary vascular complication, stroke, myocardial infarction, stent thrombosis, revascularization, death)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Nef, Prof., MD, Study Director — Herzzentrum Segeberger Kliniken GmbH
Locations (1):
- Herzzentrum Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No